CLINICAL TRIAL: NCT03624413
Title: InTSHA: Interactive Transition Support for HIV-infected Adolescents Using Social Media
Acronym: InTSHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: University of KwaZulu (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Brian Zanoni, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00116921; K23MH114771 (NIH)
Record Dates: First submitted 2018-06-13; First posted 2018-08-10 (Actual); Results first posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-09

CONDITIONS: HIV-1-infection; Adolescent Behavior
Keywords: Adolescent; HIV; Transition care; Mobile health; Social media; South Africa
MeSH Terms: conditions — Adolescent Behavior | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: A pilot randomized controlled trial with 40 adolescents receiving a social media intervention and 40 adolescents receiving standard of care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Media Intervention (Experimental): Adolescent HIV-positive participants receiving the social media intervention.
  Interventions: Behavioral: Social Media Intervention
- Standard of Care (Active Comparator): Adolescent HIV-positive participants receiving the standard of care.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Behavioral: Social Media Intervention — The social media intervention is a behavioral intervention developed by the study investigators and is delivered via mobile phones. The intervention uses the Social-ecological Model of Adolescent and Young Adult Readiness to Transition (SMART) model, highlighting modifiable targets of intervention that can be addressed through a social media platform. The SMART model incorporates modifiable factors such as knowledge, skills/self-efficacy, relationships and social support that can be targets of interventions to improve transition care. The SMART model emphasizes eight modifiable factors, three key stakeholders (adolescents, caregivers, and clinicians) and their interconnected relationship in influencing successful transition to adult care. The intervention is designed to overcome barriers and enhance facilitators to transitioning care among adolescents living with HIV who are transitioning to adult care in South Africa.
  Arms: Social Media Intervention
Other: Standard of Care — Standard of care transition from pediatric to adult care for HIV.
  Arms: Standard of Care

SUMMARY:
The goal of this study is to develop and evaluate a social media behavioral intervention based on the Social-ecological Model of Adolescent and Young Adult Readiness to Transition (SMART) to improve transition care for adolescents living with HIV in South Africa. Participants will be randomized to receive the social media intervention or the standard of care.

DETAILED DESCRIPTION:
South Africa has the highest burden of adolescents living with HIV in the world and adolescents are poorly prepared for transition from pediatric to adult services. For a large majority of South Africans living with HIV, ART was not available until 2004. This delay contributed to nearly 500,000 perinatal HIV infections in the late 1990s and early 2000s. With large scale-up and improved access to ART in recent years, survivors of perinatal HIV infection are now reaching adolescence and beyond. As the wave of perinatally HIV-infected adolescents matures, an estimated 320,000 adolescents will transfer from pediatric- or adolescent-based clinics to adult services in the next 10 years in South Africa. Currently, perinatally HIV-infected adolescents enter adult care at variable ages and developmental stages, without necessary preparation or support through the process. This study will develop and evaluate an innovative intervention designed to address this critical problem.

The SMART model incorporates modifiable factors such as knowledge, skills/self-efficacy, relationships and social support that can be targets of interventions to improve transition care. Medical care during adolescence is typically complicated by increased risk-taking behavior, as well as decreased caregiver involvement, which occur during a time of rapid physical, emotional, and cognitive development. When adolescents transition to adult care, they often do not receive the coordinated services that they received under pediatric care. Qualitative studies with adolescents and clinicians from sub-Saharan Africa suggest that peer support, collaboration with health providers, and communication between adult and pediatric providers might assist in transition to adult services. The SMART model emphasizes eight modifiable factors, three key stakeholders (adolescents, caregivers, and clinicians) and their interconnected relationship in influencing successful transition to adult care.The social media intervention for this study incorporates these stakeholders and addresses the modifiable factors in the SMART model to improve transition care for adolescents living with HIV.

Social media is defined as internet-based applications that allow the creation and exchange of user generated content. A recent meta-analysis found that social support was the most common reason for patients to use social media for health purposes. Social media has also been used to improve the relationship between caregivers and patients when switching caregivers, a major barrier to transition for adolescents in South Africa. Although results vary in different settings, a recent meta-analysis has shown overall improved adherence and viral suppression among adults living with HIV using social media based health services technology. Social media can address the modifiable variables in the SMART model such as knowledge, self-efficacy, goals, relationships, peer and social support, which could ultimately improve virologic suppression and retention in care during the transition to adult services.

The researchers will perform a pilot randomized controlled trial with 40 adolescents receiving the social media intervention and 40 adolescents receiving standard of care. In-depth interviews and quantitative surveys with adolescents living with HIV will be used to assess the acceptability and feasibility of the intervention. The secondary outcomes of peer support, connection to clinical staff, retention in care, and viral suppression will also be examined at baseline and 6 months after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Aged 15 to 19 years
* Perinatally HIV-infected
* Receiving ART for at least 6 months
* Fully aware of their HIV status

Exclusion Criteria:

* Inability to read and/or speak English or Zulu
* Severe mental or physical illness preventing informed consent

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2022-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian C Zanoni, MD, Principal Investigator — Emory University
Locations (1):
- University of Kwazulu-Natal, Westville, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be available on request and will include demographic data, age, sex, baseline cluster of differentiation 4 (CD4), viral load, results of baseline and end of study questionnaires on transition readiness, self-esteem, social support, connection to clinic and end points of acceptability, feasibility, retention in care and viral suppression.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual participant data will be made available for sharing beginning after publication of this study, with no end date.
Access Criteria: Requests for sharing the data are made by contacting Dr. Zanoni. A data sharing agreement is required before data can be accessed.

REFERENCES:
- [Derived] Zanoni BC, Archary M, Sibaya T, Goldstein M, Bergam S, Denton D, Cordero V, Peng C, Psaros C, Marconi VC, Haberer JE. Mobile Phone-Based Intervention Among Adolescents Living With Perinatally Acquired HIV Transitioning from Pediatric to Adult Care: Protocol for the Interactive Transition Support for Adolescents Living With HIV using Social Media (InTSHA) Study. JMIR Res Protoc. 2022 Jan 21;11(1):e35455. doi: 10.2196/35455. PMID 35060907

RESULTS

PARTICIPANT FLOW:
Groups:
- InTSHA Social Media Intervention: Adolescent HIV-positive participants receiving the InTSHA social media intervention.
  Social Media Intervention: The InTSHA social media intervention is a behavioral intervention developed by the study investigators and is delivered via mobile phones. The intervention uses the Social-ecological Model of Adolescent and Young Adult Readiness to Transition (SMART) model, highlighting modifiable targets of intervention that can be addressed through a social media platform. The SMART model incorporates modifiable factors such as knowledge, skills/self-efficacy, relationships and social support that can be targets of interventions to improve transition care. The SMART model emphasizes eight modifiable factors, three key stakeholders (adolescents, caregivers, and clinicians) and their interconnected relationship in influencing successful transition to adult care. The intervention is designed to overcome barriers and enhance facilitators to transitioning care among adolescents living with HIV who are transitioning to adult care in South Africa.
Period: Overall Study
Arm/Group | InTSHA Social Media Intervention | Standard of Care
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- InTSHA Social Media Intervention: Adolescent HIV-positive participants receiving the InTSHA social media intervention.
- Total: Total of all reporting groups
Arm/Group | InTSHA Social Media Intervention | Standard of Care | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.9 (1.2) | 17.0 (1.3) | 16.9 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 21 | 22 | 43
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  South Africa | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Intervention Measure Score
Description: The acceptability score is based on a validated acceptability questionnaire, the Acceptability of Intervention Measure (Proctor et al., 2011). Acceptability of the intervention is assessed with 4 questions rated on a 5-point scale, where 1 = completely disagree and 5 = completely agree. The total score is the average of item scores and ranges from 1 to 5 with higher scores indicating greater acceptability of the InTSHA intervention.
Time Frame: Month 6
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | InTSHA Social Media Intervention
Number analyzed (Participants) | 40
score on a scale | 4.1 [2.38 to 5.00]

2. Primary Outcome: Number of Participants Completing Intervention Sessions
Description: Feasibility of the intervention is reported as the number of participants randomized to the InTSHA intervention who participated in 8 to 10 sessions, 5 to 7 sessions, or fewer than 5 sessions.
Time Frame: Up to Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | InTSHA Social Media Intervention
Number analyzed (Participants) | 40
Participants
  Participated in 8 to 10 sessions | 15
  Participated in 5 to 7 sessions | 9
  Participated in less than 5 sessions | 16

3. Secondary Outcome: Change in Child and Adolescent Social Support Scale (CASSS) Score
Description: Social support from peers is assessed using 10 items of the Child and Adolescent Social Support Scale (friend support subscale). Responses are given on a 6-point scale where 1 = never and 6 = always. Total scores range from 10 to 60, where higher scores represent greater social support from peers. The change from baseline is calculated as the Month 6 score minus the Baseline score. A positive value means that the scores at Month 6 increased from what they were at Baseline.
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | InTSHA Social Media Intervention | Standard of Care
Number analyzed (Participants) | 36 | 38
score on a scale | 3.31 (9.37) | 1.74 (12.36)

4. Secondary Outcome: Change in Connection to Clinic Score
Description: A modified version of the Working Alliance Inventory is used to measure how connected participants feel to the clinical staff and medical team. Ten items are responded to on a 4-point scale where 0 = strongly disagree and 3 = strongly agree. Total scores range from 0 to 30 where higher scores indicate increased feelings of connection with clinical staff. The change from baseline is calculated as the Month 6 score minus the baseline score. A positive value means that the scores at Month 6 increased from what they were at baseline.
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | InTSHA Social Media Intervention | Standard of Care
Number analyzed (Participants) | 36 | 38
score on a scale | 0.44 (6.35) | 0.42 (5.42)

5. Secondary Outcome: Number of Participants Retained in Care
Description: Retention in care is assessed as a composite outcome of missing any pharmacy refills of antiretroviral medication and/or missing any clinic visits in the last 6 months. Participants are considered as retained in care if they did not miss any pharmacy refills or clinic visits.
Time Frame: Up to Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | InTSHA Social Media Intervention | Standard of Care
Number analyzed (Participants) | 40 | 40
Participants | 39 | 35

6. Secondary Outcome: HIV Viral Suppression
Description: HIV-1 viral load is measured in copies per milliliter (mL) and viral suppression is considered <200 copies/mL.
Time Frame: Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | InTSHA Social Media Intervention | Standard of Care
Number analyzed (Participants) | 40 | 40
Participants
  No viral suppression (>200 copies/mL) | 5 | 4
  Viral suppression (<200 copies/mL) | 35 | 36

7. Other Pre Specified Outcome: Change in Rosenberg's Self-Esteem Scale Score
Description: The Rosenberg's Self-Esteem Scale is a 10-item instrument assessing self-esteem. Responses are given on a 4-point scale where 0 = strongly disagree and 3 = strongly agree. Total scores range 0 to 30 and higher scores indicate greater self-esteem. The change in score is the Month 6 score subtracted by the Baseline score. A positive values indicates that the self-esteem score increased by the end of the study.
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | InTSHA Social Media Intervention | Standard of Care
Number analyzed (Participants) | 39 | 38
score on a scale | 0.51 (5.22) | -0.39 (5.38)

8. Other Pre Specified Outcome: Change in HIV Adolescent Readiness for Transition Scale (HARTS) Score
Description: The HIV Adolescent Readiness for Transition Scale (HARTS) includes 16 items that are responded to on a 5-point scale where 0 = no, 1 = no, but I am learning, 2 = yes, a little bit, 3 = yes, almost always, and 4 = yes, always. Total scores range from 0 to 64 and higher scores indicate greater readiness to transition to adult care. The change from baseline is calculated as the Month 6 score minus the Baseline score. A positive value means that the scores at Month 6 increased from what they were at Baseline.
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | InTSHA Social Media Intervention | Standard of Care
Number analyzed (Participants) | 39 | 38
score on a scale | 0.46 (0.79) | 0.30 (0.91)

ADVERSE EVENTS:
Time Frame: Information about adverse events was collected from the time individuals gave consent to participate through the final assessment at Month 6.
Arm/Group | InTSHA Social Media Intervention | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/13/NCT03624413/Prot_SAP_001.pdf
  • Informed Consent Form (2021-03-06): https://cdn.clinicaltrials.gov/large-docs/13/NCT03624413/ICF_000.pdf